CLINICAL TRIAL: NCT02963831
Title: A Phase 1/2 Dose Escalation Study With Expansion Cohorts to Investigate the Safety, Biologic and Anti-tumor Activity of ONCOS-102 in Combination With Durvalumab in Subjects With Advanced Peritoneal Malignancies
Brief Title: A Study to Investigate ONCOS-102 in Combination With Durvalumab in Subjects With Advanced Peritoneal Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Cancer Research Institute, New York City (Other); MedImmune LLC (Industry); Targovax ASA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2015-008
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer; Ovarian Cancer; Appendiceal Cancer
Keywords: Oncos-102; Durvalumab; Peritoneal; Cyclophosphamide
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Appendiceal Neoplasms | interventions — durvalumab; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: The Phase 1 cohorts were enrolled sequentially. In Phase 2, the two expansion cohorts are enrolled in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: ONCOS-102 Dose Escalation (Experimental): ONCOS-102, 1 x 10^11 viral particles (VPs) monotherapy for 6 weeks, followed by durvalumab 1500 mg starting on Day 71.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered intravenously (IV) 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused intraperitoneally (IP) in a total volume of 500 mL saline (0.9 mg/mL sodium chloride [NaCl] in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose every 4 weeks (Q4W) for 10 cycles, starting on Day 71.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
  Interventions: Biological: ONCOS-102; Drug: Durvalumab; Drug: Cyclophosphamide
- Cohort B: ONCOS-102 Dose Escalation (Experimental): ONCOS-102, 1 x 10^11 VPs + durvalumab 1500 mg starting on Day 15.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused IP in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose Q4W for 12 cycles, starting on Day 15.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
  Interventions: Biological: ONCOS-102; Drug: Durvalumab; Drug: Cyclophosphamide
- Cohort 1: Epithelial Ovarian Cancer (Experimental): ONCOS-102, 3 x 10^11 VPs + durvalumab 1500 mg starting on Day 15.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused IP in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose Q4W for 12 cycles, starting on Day 15.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
  Interventions: Biological: ONCOS-102; Drug: Durvalumab; Drug: Cyclophosphamide
- Cohort 2: Metastatic Colorectal Cancer (Experimental): ONCOS-102, 3 x 10^11 VPs + durvalumab 1500 mg starting on Day 15.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused IP in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose Q4W for 12 cycles, starting on Day 15.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
  Interventions: Biological: ONCOS-102; Drug: Durvalumab; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ONCOS-102 — ONCOS-102 was administered by intraperitoneal infusion at weekly intervals for 6 weeks.
  Other Names: Adenovirus Vector (Ad5/3-D24-GMCSF), Expressing GM-CSF (GM-CSF-encoding adenovirus)
Drug: Durvalumab — Durvalumab was administered by IV infusion once every four weeks for a total of 10 (Cohort A) or 12 four-week cycles.
  Other Names: MEDI4736; Imfinzi®
Drug: Cyclophosphamide — A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  Other Names: Cytoxan®

SUMMARY:
This is a two-part Phase 1/2 dose escalation and dose expansion study of an Adenovirus Vector (Ad5/3-D24-GMCSF), Expressing GM-CSF (GM-CSF-encoding adenovirus), ONCOS-102, in combination with anti-programmed death ligand-1 (PD-L1) antibody, durvalumab, in adult subjects with peritoneal disease who have failed prior standard chemotherapy and have histologically confirmed epithelial ovarian cancer or metastatic colorectal cancer.

DETAILED DESCRIPTION:
ONCOS-102 will be administered intraperitoneally (IP) at weekly intervals for 6 weeks.

A bolus dose of 300 mg cyclophosphamide (CPO) will be administered intravenously (IV) 1 to 3 days before the first infusion of ONCOS-102. Durvalumab will be administered by IV infusion once every four weeks (Q4W) for a total of 12 four-week cycles.

Phase 1 of the study is a dose escalation phase, which will use a 3+3 design to evaluate the safety of ONCOS-102 monotherapy before initiation of durvalumab and to identify the recommended combination dose (RCD) of a fixed dose of durvalumab (1500 mg) + ONCOS-102 at 2 dose levels (1 x 10^11 viral particles (VPs) and 3 x 10^11 VPs).

Subjects treated at the RCD of 3 x 10^11 VPs ONCOS-102 will be included in the Phase 2 expansion cohort based on their tumor diagnosis.

Phase 2 of the study is the dose expansion phase, which will further explore the safety and anti-tumor activity for the RCD in 2 expansion cohorts with peritoneal disease:

1. Epithelial ovarian cancer
2. Metastatic colorectal cancer

Simon's 2-Stage MINIMAX Design will be used in Phase 2 for Expansion Cohorts 1 and 2. In the first stage, 18 subjects will be enrolled in Cohort 1 and 13 subjects in Cohort 2 (including the 6 subjects at the RCD from the dose escalation phase).

If 5 or more subjects in Cohort 1, or one or more subjects in Cohort 2, demonstrate clinical benefit (defined as percentage of subjects who are not in progression at end of Week 24), 15 additional subjects will be enrolled in Stage 2 of Cohort 1, and 14 additional subjects will be enrolled in Stage 2 of Cohort 2.

The primary endpoint is the percentage of subjects who are not in progression at the end of Week 24 as measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with peritoneal disease who have failed prior standard chemotherapy and have histologic confirmation of epithelial ovarian cancer or metastatic colorectal cancer (CRC) including cancer originating from the appendix.
2. Subject is willing to undergo a core needle biopsy during screening and Cycle 2, Study Week 5. Archival tumor samples are requested but are not required for eligibility.
3. Previously treated for advanced cancer with no additional therapy options available known to prolong survival.
4. Laboratory parameters for vital functions should be in the normal range or not clinically significant.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.

Exclusion Criteria:

1. Treatment with an investigational agent within 4 weeks of starting study treatment or prior treatment with a checkpoint inhibitor (cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], programmed cell death protein 1 [PD-1] or programmed death ligand 1 [PD-L1] antibodies).
2. Subject has known active central nervous system metastasis, glioma and nervous system malignancies including carcinomatous meningitis. Subjects with asymptomatic brain metastases or spinal cord compression who have been treated, are considered stable, and who have not received corticosteroids or anticonvulsants for at least 28 days prior to screening may be included. Subject has other active malignancy.
3. Known immunodeficiency or known to have evidence of acute or chronic human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C or other uncontrolled inter-current illnesses.
4. Ongoing bowel perforation or presence of bowel fistula or abscess or history of small or large bowel obstruction within 3 months of registration, including subjects with palliative gastric drainage catheters. Subjects with palliative diverting ileostomy or colostomy are allowed if they have been symptom-free for more than 3 months.
5. Subjects with clinically significant cardiovascular disease, history of organ transplant or allogeneic bone marrow transplant, active known or history of autoimmune disease that might recur or major surgery within 28 days prior to the first dose or still recovering from prior surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Facility, San Diego, California
  - Research Facility, Miami, Florida
  - Research Facility, Buffalo, New York
  - Research Facility, New York, New York
  - Research Facility, Toledo, Ohio
  - Research Facility, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 subjects were enrolled and 64 received treatment with study therapy.
Groups:
- Cohort A: ONCOS-102 Dose Escalation: ONCOS-102, 1 x 10^11 viral particles (VPs) monotherapy for 6 weeks, followed by durvalumab 1500 mg starting on Day 71.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered intravenously (IV) 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused intraperitoneally (IP) in a total volume of 500 mL saline (0.9 mg/mL sodium chloride [NaCl] in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose every 4 weeks (Q4W) for 10 cycles, starting on Day 71.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
  .
Period: Overall Study
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Started (Started includes all subjects who received at least one dose of study therapy.) | 4 | 5 | 19 | 36
Completed (Completed includes all subjects who completed 12 cycles of treatment.) | 0 | 1 | 0 | 1
Not Completed | 4 | 4 | 19 | 35
Not completed — Progressive Disease | 3 | 3 | 16 | 27
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study medication.
Groups:
- Cohort A: ONCOS-102 Dose Escalation: ONCOS-102, 1 x 10^11 viral particles (VPs) monotherapy for 6 weeks, followed by durvalumab 1500 mg starting on Day 71.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered intravenously (IV) 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused intraperitoneally (IP) in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose every 4 weeks (Q4W) for 10 cycles, starting on Day 71.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
  .
- Cohort BL ONCOS-102 Dose Escalation: ONCOS-102, 1 x 10^11 VPs + durvalumab 1500 mg starting on Day 15.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused IP in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose Q4W for 12 cycles, starting on Day 15.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
- Total: Total of all reporting groups
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort BL ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer | Total
Number analyzed (Participants) | 4 | 5 | 19 | 36 | 64
Age, Continuous [Median (Full Range); unit: years] | 54.0 [37 to 68] | 54.0 [46 to 75] | 67.0 [49 to 77] | 58.5 [39 to 74] | 60.5 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 19 | 21 | 49
  Male | 0 | 0 | 0 | 15 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 4 | 7
  Not Hispanic or Latino | 3 | 4 | 17 | 30 | 54
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 4
  White | 2 | 4 | 16 | 32 | 54
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 19 | 36 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) and Dose Limiting Toxicities (DLTs)
Description: All Adverse events (AEs) were coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 19.0 and classified by MedDRA system organ class (SOC) and preferred term. The severity of AEs was assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03. Adverse events (AEs) were reported based on clinical laboratory tests, vital signs, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent was signed through 90 days after the last dose of study treatment. TEAEs are those that occurred or worsened after administration of the first dose of study treatment.
  Deaths within the AE Reporting Period included all deaths that occurred during the study treatment period, or up to 90 days after the administration of the last dose of study drug or initiation of a new treatment.
Time Frame: up to 31 months (90 days after the last dose of study medication).
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B ONCOS-102 Dose Escalation: ONCOS-102, 1 x 10^11 VPs + durvalumab 1500 mg starting on Day 15.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused IP in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose Q4W for 12 cycles, starting on Day 15.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 36
Participants
  Treatment-emergent Adverse Event (TEAE) | 4 | 5 | 19 | 36
  Treatment-related Adverse Event (TRAE) | 4 | 5 | 17 | 30
  Serious Adverse Event (SAE) | 3 | 3 | 9 | 22
  Treatment-related SAE | 0 | 2 | 2 | 4
  Dose-limiting Toxicity (DLT) | 0 | 0 | 0 | 0
  Death | 1 | 1 | 6 | 9
  DLTs: number analyzed (Participants) | 4 | 5 | 3 | 5
  DLTs | 0 | 0 | 0 | 0

2. Primary Outcome: Progression-free Survival (PFS) at Week 24 as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up starting 8 weeks after the last disease assessment. Per RECIST 1.1, target lesions were categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; PD: ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
  PFS was measured from the date of the first dose of study treatment to the date of earliest disease progression or to the date of death, if disease progression does not occur. Per RECIST 1.1, progressive disease (PD) is defined as a ≥ 20% increase in the sum of the longest diameter of target lesions or the development of new lesions.
Time Frame: Up to 24 weeks
Population: All subjects who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 36
Participants
  Subjects Without Progression | 0 | 1 | 0 | 2
  Subjects Who Progressed or Died | 4 | 4 | 19 | 34

3. Secondary Outcome: Median Progression-free Survival (PFS) as Measured by Response Evaluation in Solid Tumors 1.1 (RECIST 1.1) Using Kaplan-Meier Method
Description: as for outcome 2
Time Frame: Up to 29 months
Population: All subjects who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 36
months | 1.5 [1.2 to NA] — Upper limit of the confidence interval was not estimable due to insufficient number of participants with events. | 1.8 [1.4 to NA] — Upper limit of the confidence interval was not estimable due to insufficient number of participants with events. | 1.8 [1.2 to 1.9] | 1.8 [1.6 to 1.9]

4. Secondary Outcome: Objective Response Rate as Measured by as Measured by Response Evaluation in Solid Tumors 1.1 (RECIST 1.1)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST 1.1 at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up starting 8 weeks after the last disease assessment. Per RECIST 1.1, target lesions were categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; PD: ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 15 months
Population: All subjects who received at least one dose of study medication and had a baseline and at least one post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 31
Participants
  CR | 0 | 0 | 0 | 0
  PR | 0 | 1 | 0 | 0
  SD | 0 | 1 | 4 | 9
  PD | 4 | 3 | 15 | 22

5. Secondary Outcome: Progression-free Survival (PFS) at Week 24 as Measured by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up starting 8 weeks after the last disease assessment. Per irRECIST, measurable lesions were categorized as follows: immune-related complete response (irCR): Complete disappearance of all target lesions; immune-related partial response (irPR): ≥ 30% decrease from baseline in the Total Measurable Tumor Burden (TMTB); immune-related progressive disease (irPD): ≥ 20% increase from nadir in TMTB; immune-related stable disease (irSD): not meeting above criteria.
  PFS was measured from the date of the first dose of study treatment to the date of earliest disease progression or to the date of death, if disease progression does not occur. Per irRECIST, irPD is defined as a ≥ 20% increase from nadir in the TMTB.
Time Frame: Up to 24 Weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 18 | 32
Participants
  Subjects Without Progression | 0 | 1 | 0 | 3
  Subjects Who Progressed or Died | 4 | 4 | 18 | 29

6. Secondary Outcome: Median Progression-free Survival (PFS) by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) as Estimated Using the Kaplan-Meier Method
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5,7, 9, and 11 during study treatment, and during on-study follow-up starting 8 weeks after the last disease assessment. Per irRECIST, measurable lesions were categorized as follows: immune-related complete response (irCR): Complete disappearance of all target lesions; immune-related partial response (irPR): ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); immune-related progressive disease (irPD): ≥ 20% increase from nadir in TMTB; immune-related stable disease (irSD): not meeting above criteria.
  PFS was measured from the date of the first dose of study treatment to the date of earliest disease progression or to the date of death, if disease progression does not occur. Per irRECIST, irPD is defined as a ≥ 20% increase from nadir in the TMTB.
Time Frame: Up to 39 months
Population: All subjects who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 36
months | 1.5 [1.2 to NA] — Upper limit of the confidence interval was not estimable due to insufficient number of participants with events. | 1.8 [1.4 to NA] — Upper limit of the confidence interval was not estimable due to insufficient number of participants with events. | 1.8 [1.2 to 1.9] | 1.9 [1.6 to 2.0]

7. Secondary Outcome: Objective Response Rate as Measured by Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), at cycles 3, 5, 7, 9, and 11 during study treatment, and during on-study follow-up starting 8 weeks after the last disease assessment. Per irRECIST, measurable lesions were categorized as follows: immune-related complete response (irCR): Complete disappearance of all target lesions; immune-related partial response (irPR): ≥ 30% decrease from baseline in the total measurable tumor burden (TMTB); immune-related progressive disease (irPD): ≥ 20% increase from nadir in TMTB; immune-related stable disease (irSD): not meeting above criteria.
Time Frame: Up to 15 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Colorectal Cancer: ONCOS-102, 3 x 10^11 VPs + durvalumab 1500 mg starting on Day 15.
  A bolus dose of 300 mg cyclophosphamide (CPO) was administered IV 1 to 3 days before the first infusion of ONCOS-102.
  ONCOS-102 was infused IP in a total volume of 500 mL saline (0.9 mg/mL NaCl in water for injection) by gravity feed or per institutional procedures for IP infusions. ONCOS-102 was to be administered weekly for a total of 6 weeks, starting on Day 1.
  Durvalumab was administered as an intravenous (IV) infusion at a fixed dose of 1500 mg in either 0.9% (w/v) saline or dextrose Q4W for 12 cycles, starting on Day 15.
  Optional durvalumab treatment extension beyond the initial 12-cycle treatment period was allowed for subjects who complete the 12-cycle treatment period with Stable Disease or better.
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 31
Participants
  irCR | 0 | 0 | 0 | 0
  irPR | 0 | 1 | 0 | 0
  irSD | 0 | 1 | 4 | 11
  irPD | 4 | 3 | 15 | 20

8. Secondary Outcome: Median Overall Survival (OS) as Estimated Using the Kaplan-Meier Method
Description: After completion of treatment, all subjects were followed for survival every 6 months up to 3 years following initiation of study treatment or until June 25, 2022 when all post-study follow-up was completed. OS was measured from the date of the first dose of study treatment to the date of death or last follow-up (June 25, 2022 when the last follow-up data was collected or earlier). Subjects lost to follow-up are censored on the date when they were last known to be alive.
Time Frame: Up to 39 months
Population: All subjects who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B: ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
Number analyzed (Participants) | 4 | 5 | 19 | 36
months | 5.9 [3.9 to NA] — Upper limit of the confidence interval was not estimable due to insufficient number of participants with events. | 10.1 [3.1 to NA] — Upper limit of the confidence interval was not estimable due to insufficient number of participants with events. | 6.6 [3.6 to 18.8] | 7.1 [4.9 to 11.5]

ADVERSE EVENTS:
Time Frame: AEs were collected up to 31 months (90 days after the last dose of study medication). All AEs occurring between the signing of informed consent and the off-study date (i.e., through 90 days after the last dose of study treatment) are documented, regardless of a causal relationship to study drug. All-cause mortality includes all deaths which were reported up for up to 39 months.
Description: AEs that occur or worsen in severity after the first dose of study treatment are considered treatment emergent (i.e., TEAEs). AE documentation includes onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Cohort A: ONCOS-102 Dose Escalation | Cohort B ONCOS-102 Dose Escalation | Cohort 1: Epithelial Ovarian Cancer | Cohort 2: Metastatic Colorectal Cancer
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/5 | 16/19 | 28/36
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/5 | 9/19 | 22/36
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 19/19 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: ONCOS-102 Dose Escalation (N=4) | Cohort B ONCOS-102 Dose Escalation (N=5) | Cohort 1: Epithelial Ovarian Cancer (N=19) | Cohort 2: Metastatic Colorectal Cancer (N=36)
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 3
Infusion site erythema (General disorders) | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Blood culture positive (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 6 | 9
Metastases to the ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: ONCOS-102 Dose Escalation (N=4) | Cohort B ONCOS-102 Dose Escalation (N=5) | Cohort 1: Epithelial Ovarian Cancer (N=19) | Cohort 2: Metastatic Colorectal Cancer (N=36)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 12 | 21
Vomiting (Gastrointestinal disorders) | 2 | 4 | 11 | 15
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 6 | 16
Constipation (Gastrointestinal disorders) | 1 | 2 | 5 | 13
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 7 | 9
Abdominal distention (Gastrointestinal disorders) | 2 | 1 | 7 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 4 | 14 | 20
Fatigue (General disorders) | 3 | 3 | 12 | 19
Chills (General disorders) | 4 | 3 | 7 | 18
Oedema peripheral (General disorders) | 1 | 1 | 1 | 4
Pain (General disorders) | 1 | 2 | 1 | 2
Influenza like illness (General disorders) | 0 | 0 | 2 | 2
Malaise (General disorders) | 2 | 0 | 0 | 2
Catheter site pain (General disorders) | 0 | 0 | 1 | 2
Oedema (General disorders) | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Complication associated with device (General disorders) | 0 | 0 | 0 | 1
Early satiety (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 1 | 0
Infusion site rash (General disorders) | 0 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0 | 0
Medical device site discharge (General disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 4 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 4
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Carbohydrate antigen 125 increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 3
Depression (Psychiatric disorders) | 0 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT02963831/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT02963831/SAP_001.pdf